CLINICAL TRIAL: NCT05981248
Title: Experiential Avoidance as the Mechanism of Mindfulness Based Intervention in Reducing Emotional Distress: Daily Dairy Research
Brief Title: Experiential Avoidance as the Mechanism of Mindfulness Intervention in Reducing Emotional Distress: Daily Dairy Research
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Peking University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: E20230815
Record Dates: First submitted 2023-08-01; First posted 2023-08-08 (Actual); Last update posted 2023-08-08 (Actual); Status verified 2023-07

CONDITIONS: Emotional Distress

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- the MIED+TAU group (Experimental): provide standard audio instructions for mindfulness exercises, introduce the nature and law of anxiety, depression and other emotions, the source of anxiety, depression and other emotional distress, and the strategies and methods to alleviate emotional distress. These exercises, knowledge and strategies are based on the latest progress in the field of psychological counseling and treatment, and their application in daily life can help alleviate anxiety, depression and other emotional problems.
  Interventions: Behavioral: Mindfulness Intervention for Emotional Distress
- the TAU-only group (No Intervention): treated as usual

INTERVENTIONS:
Behavioral: Mindfulness Intervention for Emotional Distress — Mindfulness Intervention for Emotional Distress (MIED) program provide standard audio instructions for mindfulness exercises, introduce the nature and law of anxiety, depression and other emotions, the source of anxiety, depression and other emotional distress, and the strategies and methods to alleviate emotional distress. These exercises, knowledge and strategies are based on the latest progress in the field of psychological counseling and treatment, and their application in daily life can help alleviate anxiety, depression and other emotional problems.
  Arms: the MIED+TAU group

SUMMARY:
This study hopes to:

1. explore whether three weeks of MIED could promote experiential avoidance.
2. explore experiential avoidance could be a mediation of outcomes of MIED.

DETAILED DESCRIPTION:
Experiential avoidance refers to individuals resisting experiences or trying to eliminate certain experiences (such as emotions, thoughts, physical feelings, memory and behavioral tendencies, etc.), and trying to adopt corresponding strategies to change these experiences and the situations in which the experiences are generated (Hayes, Wilson, Gifford, Follette, & Strosahl, 1996). Experiential avoidance has been proved to be a maintenance factor for many psychological disorders (Boelen & Reijntjes, 2008), and trying to hide or suppress unpleasant thoughts, feelings and physical feelings will increase the frequency and pain of these same experiences (Gross,1998; Gross,2002; Sloan, 2004; Wegner, 1994). According to some reviews, experiential avoidance is one of the beneficial effects of mindfulness (Brown, Bravo, Roos, & Pearson, 2015; Shapiro et al., 2006). However, no study has examined experiential avoidance as mediator in mindfulness intervention whether in the between-subject or in within-subject level . Therefore, this study uses daily diary research explore the role of experiential avoidance as the effective mechanism of mindfulness intervention.

ELIGIBILITY:
Inclusion Criteria:

* Subjects with scores greater than 21 on the Kessler Psychological Distress Scale.

Exclusion Criteria:

* Subjects who could not access the Internet;
* Subjects with insufficient Chinese ability;
* Subjects who have participated in mindfulness based projects for more than 6 weeks before, and / or the current frequency of meditation practice is more than once a week;
* Patients with schizophrenia or psychotic affective disorder, current organic mental disorder, substance abuse disorder and generalized developmental disorder;
* Subjects at risk of suicide.

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 200 (Estimated)
Dates: Start 2023-08-15 (Estimated); Primary Completion 2023-11-30 (Estimated); Study Completion 2023-11-30 (Estimated)

PRIMARY OUTCOMES:
Weekly changes of Five Facet Mindfulness Questionnaire during the intervention | pre-intervention; weekly during the 7-week intervention; after the 7-week intervention
  The Five Facet Mindfulness Questionnaire is a self-reported questionnaire measuring mindfulness levels. Scores range from 39 to 195, with higher scores indicating higher levels of mindfulness.
Weekly changes of Chinese Perceived Stress Scale during the intervention | pre-intervention; weekly during the 7-week intervention; after the 7-week intervention
  The Chinese Perceived Stress Scale is a self-reported questionnaire measuring stress. Scores range from 0 to 56, with higher scores indicating higher levels of stress.
Weekly changes of 10-item Kessler Psychological Distress Scale during the intervention | pre-intervention; weekly during the 7-week intervention; after the 7-week intervention
  The 10-item Kessler Psychological Distress Scale is a self-reported questionnaire measuring distress. Scores range from 10 to 50, with higher scores indicating higher levels of distress.
Weekly changes of Overall Anxiety Severity and Impairment Scale during the intervention | pre-intervention; weekly during the 7-week intervention; after the 7-week intervention
  The Overall Anxiety Severity and Impairment Scale is a self-reported questionnaire measuring anxiety. Scores range from 0 to 20, with higher scores indicating higher levels of anxiety.
Weekly changes of Overall Depression Severity and Impairment Scale during the intervention | pre-intervention; weekly during the 7-week intervention; after the 7-week intervention
  The Overall Depression Severity and Impairment Scale is a self-reported questionnaire measuring depression. Scores range from 0 to 20, with higher scores indicating higher levels of depression.
Weekly changes of Inner Peace Scale during the intervention | pre-intervention; weekly during the 7-week intervention; after the 7-week intervention
  The Inner Peace Scale is a self-reported questionnaire measuring peace. Scores range from 0 to 28, with higher scores indicating higher levels of peace.
Weekly changes of Depression-Anxiety-Stress Scale during the intervention | pre-intervention; weekly during the 7-week intervention; after the 7-week intervention
  The Depression-Anxiety-Stress Scale is a self-reported questionnaire measuring psychological health. Scores range from 0 to 63, with higher scores indicating higher levels of depression, anxiety or stress.
Weekly changes of Acceptance and Action Questionnaire-II during the intervention | pre-intervention; weekly during the 7-week intervention; after the 7-week intervention
  The Acceptance and Action Questionnaire-II is a self-reported questionnaire measuring experiential avoidance. Scores range from 7 to 49, with higher scores indicating higher levels of experiential avoidance.
Weekly changes of Brief Experiential Avoidance Questionnaire during the I intervention | pre-intervention; weekly during the 7-week intervention; after the 7-week intervention
  The Brief Experiential Avoidance Questionnaire is a self-reported questionnaire measuring experiential avoidance. Scores range from 15 to 90, with higher scores indicating higher levels of experiential avoidance.
Daily changes of experiential avoidance | once a day in the first three weeks of the intervention
  There are 7 items, 4 of which evaluate the use of specific experiential avoidance strategies today, including distraction , redundant thinking, thought suppression and reassessment and 3 of which evaluate today's broader experiential avoidance. Scores range from 7 to 35, with higher scores indicating higher levels of experiential avoidance.
Daily changes of anxiety | once a day in the first three weeks of the intervention
  Daily anxiety was assessed using a 6-item shortened version of the State-Trait Anxiety Inventory. Scores range from 6 to 24, with higher scores indicating higher levels of anxiety.
Daily changes of depression | once a day in the first three weeks of the intervention
  Daily depressive symptoms were measured by a 10-item modified version of the Centre for Epidemiologic Studies Depressive Scale with item wordings adapted to include the word 'today' and the instructions modified. Scores range from 0 to 30, with higher scores indicating higher levels of depression.
Daily changes of positive and negative affect | once a day in the first three weeks of the intervention
  Daily positive and negative affect were measured using the 10-itemInternational Positive and Negative Affect Schedule-Short Form Scale. Scores range from 5 to 25, with higher scores indicating higher levels of positive/negative affect.
Daily stressor exposure | once a day in the first three weeks of the intervention
  Daily stressor exposure was measured using a 7-item scale from the Daily Inventory of Stressful Events. if at least one stressor event was experienced by the participant within the day, it was then categorized as a stressor day. If no stressor events were experienced on the day, it was categorized as a non-stressor day.
Daily mindfulness | once a day in the first three weeks of the intervention
  5 items with the highest factor from each subscale of the Five-Facet Mindfulness Questionnaire were chosen. Scores range from 5 to 25, with higher scores indicating higher levels of mindfulness.

CONTACTS AND LOCATIONS:
Overall Officials: Xinghua Liu, Principal Investigator — School of Psychological and Cognitive Sciences, Peking University

IPD SHARING:
Plan to Share IPD: No